CLINICAL TRIAL: NCT05819827
Title: Investigation of Associations Between Chemotherapy-Induced Nausea in Patients With Genitourinary, Sarcoma or Melanoma Cancers and Changes in Gut Microbiome: Potential for Precision Therapeutics
Brief Title: Associations Between Chemotherapy-Induced Nausea in Patients With Genitourinary, Sarcoma or Melanoma Cancers and Changes in Gut Microbiome: Potential for Precision Therapeutics
Status: Terminated | Type: Observational
Why Stopped: Low/slow accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Komal P. Singh, Principal Investigator, Mayo Clinic
Other Study IDs: 22-010340; NCI-2023-02454 (Registry Identifier: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Bladder Cancer; Prostate Cancer; Testicular Cancer; Bladder Carcinoma; Genitourinary System Carcinoma; Malignant Testicular Neoplasm; Melanoma; Prostate Carcinoma; Sarcoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Prostatic Neoplasms; Testicular Neoplasms; Melanoma; Sarcoma | interventions — Blood Specimen Collection; Histocompatibility Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients will collect stool for microbiome analysis at baseline (i.e., 3 +2 days prior to chemotherapy) and again 5-7 days following initiation of chemotherapy.
  Blood samples will be collected prior to their first chemotherapy treatment, and in the second week after chemotherapy. The blood sample will be used for several assays that include gene expression, immune cell profiling, metabolite analytics, and additional omics assays.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with genitourinary cancers: Genitourinary medical oncologists and study coordinators will identify patients with genitourinary cancers (i.e., bladder cancer, prostate cancer, and testicular cancer) who will receive moderate to high emetogenic chemotherapy regimen.
  Interventions: Other: Blood and Tissue

INTERVENTIONS:
Other: Blood and Tissue — Patients will collect stool for microbiome analysis at baseline (i.e., 3 +2 days prior to chemotherapy) and again 5-7 days following initiation of chemotherapy.
  Blood samples will be collected prior to their first chemotherapy treatment, and in the second week after chemotherapy.

SUMMARY:
The objective of this pilot cohort study is to investigate associations between CIN and changes in gut microbiome composition profiles.

DETAILED DESCRIPTION:
The long-term goal of this study is to alleviate the occurrence of CIN and to improve chemotherapy treatment outcomes. The identification of associations between CIN and chemotherapy-induced changes in gut microbiome composition profiles will increase our understanding of these mechanisms that underlie CIN. An increased understanding of the underlying mechanisms will provide targets for the development of novel interventions to help alleviate CIN.

ELIGIBILITY:
Inclusion Criteria:

* at least 20 years of age
* last chemotherapy more than 3 years ago
* scheduled to receive either moderate to highly emetogenic chemotherapy with or without targeted therapies including immunotherapies) or immunotherapies/targeted therapies alone that can lead to toxicity symptoms for example, nausea and fatigue.
* Patients receiving chemotherapy and/or immunotherapy treatment at a Mayo Clinic infusion center or an infusion center outside of Mayo Clinic

Exclusion Criteria:

* concurrent radiation therapy
* concurrent antibiotic treatment
* concurrent oncolytic virus treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a diagnosis of bladder cancer, prostate cancer, testicular cancer, cancerous sarcoma and melanoma- planning to receive moderate to highly emetogenic chemotherapy will be recruited at Mayo Clinic, Arizona, Mayo Clinic Rochester, MN and Mayo Clinic Florida.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Change in patient recruitment | Baseline, 14 days
  Evaluate the feasibility of patient recruitment by using descriptive statistics to determine number of patients approached and number of patients enrolled.
Change in patient retention | Baseline, 14 days
  Evaluate the feasibility of patient retention by using descriptive statistics to determine number of patients who completed the questionnaires at both assessments.
Change in patient specimen collection | Baseline, 14 days
  Evaluate the feasibility of patient specimen collection by using descriptive statistics to determine number patients who provided stool samples at both assessments.
Change of the gut microbiome | Up to 10 months
  Evaluate for changes in alpha and beta diversity as well as composition of the gut microbiome pre- and post-chemotherapy in patients who do and do not report chemotherapy-induced nausea (CIN) after chemotherapy. Region V3-V5 of the 16s rRNA gene will be targeted for sequencing and submitted to trimmomatic for reads trimming and quality control.
Associations between microbial composition functional profiles | Up to 10 months
  Examine associations between microbial composition functional profiles pre- and post-chemotherapy in patients who report chemotherapy-induced nausea (CIN) after chemotherapy. Change in relative abundance of genus associated with CIN occurrence will be used to predict the function of the genus. We will use PiCrust to perform functional profiling.
Evaluate for differentially abundant metabolites | Up to 10 months
  Evaluate for differentially abundant metabolites associated with microbiome diversity in patients who do and do not report chemotherapy-induced nausea (CIN) after chemotherapy. Metabolomics profiling of stool samples pre- and post-chemotherapy using liquid chromatography-tandem mass spectrometry (LC-MS/MS).
Evaluate for perturbed metabolic pathways | Up to 10 months
  Evaluate for perturbed metabolic pathways associated with microbiome diversity in patients who do and do not report chemotherapy-induced nausea (CIN) after chemotherapy. Metabolomics profiling will be performed on stool samples pre- and post-chemotherapy using liquid chromatography-tandem mass spectrometry (LC-MS/MS), as well as RNA-Seq analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Komal P. Singh, Ph.D., R.N., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials